CLINICAL TRIAL: NCT05687422
Title: A Randomized Controlled Study of Two Patterns of Micropulse Laser in the Treatment of Chronic Central Serous Chorioretinopathy
Brief Title: Two Patterns of Micropulse Laser in the Treatment of Chronic Central Serous Chorioretinopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Hospital (Other Government)
Responsible Party: Principal Investigator, Yu Xiaobing, Prof., Beijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-I2M-C&T-B-093
Record Dates: First submitted 2022-12-25; First posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Central Serous Chorioretinopathy
MeSH Terms: conditions — Central Serous Chorioretinopathy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 100μm laser spot diameter group (Experimental)
  Interventions: Procedure: 100μm laser spot diameter micropulse laser
- 200μm laser spot diameter group (Active Comparator)
  Interventions: Procedure: 200μm laser spot diameter micropulse laser

INTERVENTIONS:
Procedure: 100μm laser spot diameter micropulse laser — 100μm laser spot diameter micropulse laser at baseline, then follow-up for 6 months
  Arms: 100μm laser spot diameter group
Procedure: 200μm laser spot diameter micropulse laser — 200μm laser spot diameter micropulse laser at baseline, then follow-up for 6 months
  Arms: 200μm laser spot diameter group

SUMMARY:
Central serous chorioretinopathy (CSC) is a common eye disease mainly involving the macular area, causing central visual acuity loss. Recently, subthreshold micropulse laser used in treating chronic CSC is proved to be safe and effective. However, some studies indicate that it's less effective than half dose photodynamic therapy (PDT). Certain physicians, including us, think that this may be related to micropulse laser parameters. Thus we need to explore better laser patterns to replace PDT in treating chronic CSC. The aim of this study is to compare the treatment effect of two different patterns of laser parameters (small and regular spot diameter) in treating chronic CSC. In this randomized, double blinded, controlled trial, by comparing the subretinal fluid regression ratio, central retinal thickness, macular microvisual field, macular vascular density, chroidal volume changes and visual acuity of two groups 6 months after micropulse laser treatment, we aim to evaluate the safety and efficacy of refined micropulse laser in treating chronic CSC.

ELIGIBILITY:
Inclusion Criteria:

* Patients age range 18-50 years
* Patients diagnosed with chronic Central serous chorioretinopathy
* Patients have signed informed consent

Exclusion Criteria:

* A history of other fundus diseases or refractive media opacity
* Patients have underwent other treatment methods for chronic Central serous chorioretinopathy
* Diopter>-6D
* A history of system diseases such as hypertension or diabetes
* A history of using local or systemic corticosteroids

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Subretinal fluid regression ratio | 6 months
  Comparing the subretinal fluid regression ratio of two groups at 6 months follow-up
Central retinal thickness changes | 6 months
  Comparing the central retinal thickness changes of two groups at 6 months

REFERENCES:
- [Derived] Zhang Y, Wang J, Liu J, Gu X, Song S, Yu X. Three-dimensional choroidal characteristics in different subtypes of central serous chorioretinopathy using swept-source optical coherence tomography angiography. Graefes Arch Clin Exp Ophthalmol. 2025 Mar;263(3):689-697. doi: 10.1007/s00417-024-06691-8. Epub 2024 Nov 19. PMID 39557692